CLINICAL TRIAL: NCT00838916
Title: A Randomized, Open-label, Parallel-group, Multicenter Study to Determine the Efficacy and Long-term Safety of Albiglutide Compared With Insulin in Subjects With Type 2 Diabetes Mellitus.
Brief Title: A Study to Determine the Safety and Efficacy of Albiglutide in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112754
Record Dates: First submitted 2009-02-05; First posted 2009-02-09 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — rGLP-1 protein; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- albiglutide weekly injection (Experimental): albiglutide weekly subcutaneous injection
  Interventions: Biological: albiglutide
- insulin glargine (Active Comparator): insulin glargine daily injection
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Biological: albiglutide — albiglutide weekly injection
  Arms: albiglutide weekly injection
Drug: insulin glargine — insulin glargine
  Arms: insulin glargine

SUMMARY:
A study to determine the safety and efficacy of albiglutide in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* BMI 20-45kg/m2 inclusive

Exclusion Criteria:

* females who are pregnant, lactating or within <6 weeks post-partum
* current symptomatic heart failure (NYHA Class III-IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 779 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (277):
- United States (255):
  - GSK Investigational Site, Alabaster, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Hueytown, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Green Valley, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Bull Shoals, Arkansas
  - GSK Investigational Site, Harrisburg, Arkansas
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Searcy, Arkansas
  - GSK Investigational Site, Buena Park, California
  - GSK Investigational Site, Cathedral City, California
  - GSK Investigational Site, Chino, California
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Commerce, California
  - GSK Investigational Site, Escondido, California
  - GSK Investigational Site, Foothill Ranch, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Lakewood, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Alamitos, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Palm Desert, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Satna Monica, California
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Tustin, California
  - GSK Investigational Site, Victorville, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Britain, Connecticut
  - GSK Investigational Site, Trumbull, Connecticut
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Middletown, Delaware
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Cocoa, Florida
  - GSK Investigational Site, Cutler Bay, Florida
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, Delray Beach, Florida
  - GSK Investigational Site, Edgewater, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Lauderdale Lakes, Florida
  - GSK Investigational Site, Marianna, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Oviedo, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Ponte Verda, Florida
  - GSK Investigational Site, Saint Cloud, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Blue Ridge, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Snellville, Georgia
  - GSK Investigational Site, Stone Mountain, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Aurora, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evergreen Park, Illinois
  - GSK Investigational Site, Gurnee, Illinois
  - GSK Investigational Site, La Grange, Illinois
  - GSK Investigational Site, Naperville, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Fishers, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, La Porte, Indiana
  - GSK Investigational Site, Lafayette, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Dubuque, Iowa
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Waterloo, Iowa
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Mission, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Fort Mitchell, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Madisonville, Kentucky
  - GSK Investigational Site, Paducah, Kentucky
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Lake Charles, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Hyattsville, Maryland
  - GSK Investigational Site, Oxon Hill, Maryland
  - GSK Investigational Site, Haverhill, Massachusetts
  - GSK Investigational Site, Bay City, Michigan
  - GSK Investigational Site, Benzonia, Michigan
  - GSK Investigational Site, Bloomfield Hills, Michigan
  - GSK Investigational Site, Cadillac, Michigan
  - GSK Investigational Site, Dearborn, Michigan
  - GSK Investigational Site, Interlochen, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Saint Clair Shores, Michigan
  - GSK Investigational Site, Brooklyn Center, Minnesota
  - GSK Investigational Site, Gulfport, Mississippi
  - GSK Investigational Site, Picayune, Mississippi
  - GSK Investigational Site, Rolling Fork, Mississippi
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, West Plains, Missouri
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Great Falls, Montana
  - GSK Investigational Site, Broken Bow, Nebraska
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Berlin, New Jersey
  - GSK Investigational Site, Elizabeth, New Jersey
  - GSK Investigational Site, Haddon Heights, New Jersey
  - GSK Investigational Site, Hainesport, New Jersey
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Stratford, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, North Massapequa, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Burlington, North Carolina
  - GSK Investigational Site, Calabash, North Carolina
  - GSK Investigational Site, Fayetteville, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Lenoir, North Carolina
  - GSK Investigational Site, Mint Hill, North Carolina
  - GSK Investigational Site, Morehead City, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Tabor City, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Canal Fulton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Mason, Ohio
  - GSK Investigational Site, Maumee, Ohio
  - GSK Investigational Site, Thornville, Ohio
  - GSK Investigational Site, Zanesville, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Ashland, Oregon
  - GSK Investigational Site, Bensalem, Pennsylvania
  - GSK Investigational Site, Carlisle, Pennsylvania
  - GSK Investigational Site, Downington, Pennsylvania
  - GSK Investigational Site, Harrisburg, Pennsylvania
  - GSK Investigational Site, Landsdale, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Tipton, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Manning, South Carolina
  - GSK Investigational Site, Murrells Inlet, South Carolina
  - GSK Investigational Site, North Myrtle Beach, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Taylors, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Columbia, Tennessee
  - GSK Investigational Site, Fayetteville, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, McKenzie, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Tullahoma, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Bedford, Texas
  - GSK Investigational Site, Cleburne, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Deer Park, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Hurst, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Lake Jackson, Texas
  - GSK Investigational Site, Lewisville, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, North Richland Hills, Texas
  - GSK Investigational Site, Odessa, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Schertz, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Sugarland, Texas
  - GSK Investigational Site, Bountiful, Utah
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, West Valley City, Utah
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Manassas, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Suffolk, Virginia
  - GSK Investigational Site, Weber City, Virginia
  - GSK Investigational Site, Renton, Washington
  - GSK Investigational Site, Richland, Washington
  - GSK Investigational Site, Selah, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Lewisburg, West Virginia
  - GSK Investigational Site, Milwaukee, Wisconsin
- Russia (6):
  - GSK Investigational Site, Arkhangelsk
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Yaroslavl
- South Africa (10):
  - GSK Investigational Site, Port Elizabeth, Eastern Cape
  - GSK Investigational Site, Johannesburg, Gauteng
  - GSK Investigational Site, Lenasia, Gauteng
  - GSK Investigational Site, Parktown, Gauteng
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Phoenix, KwaZulu-Natal
  - GSK Investigational Site, Somerset West, Western Province
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Kempton Park
  - GSK Investigational Site, Parow
- United Kingdom (6):
  - GSK Investigational Site, Blackpool, Lancashire
  - GSK Investigational Site, Sunbury-on-Thames, Middlesex
  - GSK Investigational Site, Port Glasgow, Renfrewshire
  - GSK Investigational Site, Coventry, West Midlands
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Home PD, Ahren B, Reusch JEB, Rendell M, Weissman PN, Cirkel DT, Miller D, Ambery P, Carr MC, Nauck MA. Three-year data from 5 HARMONY phase 3 clinical trials of albiglutide in type 2 diabetes mellitus: Long-term efficacy with or without rescue therapy. Diabetes Res Clin Pract. 2017 Sep;131:49-60. doi: 10.1016/j.diabres.2017.06.013. Epub 2017 Jun 15. PMID 28683300
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- [Derived] Weissman PN, Carr MC, Ye J, Cirkel DT, Stewart M, Perry C, Pratley R. HARMONY 4: randomised clinical trial comparing once-weekly albiglutide and insulin glargine in patients with type 2 diabetes inadequately controlled with metformin with or without sulfonylurea. Diabetologia. 2014 Dec;57(12):2475-84. doi: 10.1007/s00125-014-3360-3. Epub 2014 Sep 11. PMID 25208756
- [Derived] Young MA, Wald JA, Matthews JE, Yang F, Reinhardt RR. Effect of renal impairment on the pharmacokinetics, efficacy, and safety of albiglutide. Postgrad Med. 2014 May;126(3):35-46. doi: 10.3810/pgm.2014.05.2754. PMID 24918790
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 112754 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112754 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112754 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112754 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112754 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112754 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112754 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) who met eligibility criteria and completed a 4 week Run-in/Stabilization Period were then randomized to a 156-week Treatment Period, followed by 8 weeks of post-treatment follow-up. A total of 1060 par. were screened; 779 par. were randomized, and 745 par. received >=1 treatment dose.
Groups:
- Albiglutide 30 mg + Metformin +/- Sulfonylurea: Participants received albiglutide 30 milligrams (mg) weekly (with up-titration to 50 mg weekly if required) as a subcutaneous injection via a fully disposable pen injector system plus metformin >=1500 mg daily plus or minus sulfonylurea from Baseline to Week 156. All participants returned for the 8-week post-treatment Follow-up Period.
- Insulin Glargine 10 Units + Metformin +/- Sulfonylurea: Participants received 10 units of insulin glargine daily (with dose adjusted weekly depending on the need for additional glycemic control) as a subcutaneous injection via a fully disposable pen injector system plus metformin >=1500 mg daily plus or minus sulfonylurea from Baseline to Week 156. All participants returned for the 8-week post-treatment Follow-up Period.
Period: Treatment Period (156 Weeks)
Arm/Group | Albiglutide 30 mg + Metformin +/- Sulfonylurea | Insulin Glargine 10 Units + Metformin +/- Sulfonylurea
Started | 504 | 241
Completed | 308 | 164
Not Completed | 196 | 77
Not completed — Adverse Event | 50 | 11
Not completed — Protocol Violation | 12 | 3
Not completed — Noncompliance | 21 | 14
Not completed — Severe or Repeated Hypoglycaemia | 1 | 0
Not completed — Lost to Follow-up | 19 | 18
Not completed — Withdrawal by Subject | 81 | 29
Not completed — Physician Decision | 6 | 1
Not completed — Termination of Study/Site by GSK | 1 | 0
Not completed — Missing | 3 | 1
Not completed — Pregnancy | 2 | 0
Period: Follow-up Period (8 Weeks)
Arm/Group | Albiglutide 30 mg + Metformin +/- Sulfonylurea | Insulin Glargine 10 Units + Metformin +/- Sulfonylurea
Started | 504 (Participants withdrawing from the Treatment Period entered the Follow-up Period.) | 241 (Participants withdrawing from the Treatment Period entered the Follow-up Period.)
Completed | 408 | 190
Not Completed | 96 | 51
Not completed — Adverse Event | 10 | 5
Not completed — Noncompliance | 6 | 5
Not completed — Lost to Follow-up | 38 | 22
Not completed — Did not Enter Follow-up Period | 7 | 7
Not completed — Withdrawn from Follow-up Participation | 26 | 12
Not completed — Physician Decision | 2 | 0
Not completed — Termination of Study/Site by GSK | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Missing | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Albiglutide 30 mg + Metformin +/- Sulfonylurea | Insulin Glargine 10 Units + Metformin +/- Sulfonylurea | Total
Number analyzed (Participants) | 504 | 241 | 745
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.8 (9.33) | 54.7 (9.75) | 55.5 (9.48)
Gender [Count of Participants; unit: Participants]
  Female | 218 | 109 | 327
  Male | 286 | 132 | 418
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 130 | 64 | 194
  American Indian or Alaskan Native | 3 | 1 | 4
  Asian - Central/South Asian Heritage | 7 | 5 | 12
  Asian - East Asian Heritage | 2 | 1 | 3
  Asian - Japanese Heritage | 0 | 1 | 1
  Asian - South East Asian Heritage | 16 | 8 | 24
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White - Arabic/North African Heritage | 7 | 2 | 9
  White - White/Caucasian/European Heritage | 342 | 158 | 500
  Other - Central American Indian | 1 | 0 | 1
  Other - Hispanic | 0 | 1 | 1
  Other - Mexican | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Glycosylated Hemoglobin (HbA1c) at Week 52
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The BL HbA1c value is defined as the last non-missing value before the start of treatment. Change from BL was calculated as the value at Week 52 minus the value at BL. Based on analysis of covariance (ANCOVA): change = treatment + BL HbA1c + prior myocardial infarction history + age category + region + current antidiabetic therapy. Difference of least squares means (albiglutide - insulin glargine) is from the ANCOVA model. The last observation carried forward (LOCF) method was used to impute missing post-Baseline HbA1c values; the last non-missing post-BL on-treatment measurement was used to impute the missing measurement. HbA1c values obtained after hyperglycemic rescue were treated as missing and were replaced with pre-rescue values.
Time Frame: Baseline and Week 52
Population: Intent-to-Treat (ITT) Population with LOCF: all randomized par. who received >=1 dose of study medication and who had a BL assessment and >=1 post-BL assessment of HbA1c. Only par. with a value at BL and at the specified visit were analyzed. Values were carried forward for par. who were rescued or discontinued from active treatment before Week 52.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c in the blood
Arm/Group | Albiglutide 30 mg + Metformin +/- Sulfonylurea | Insulin Glargine 10 Units + Metformin +/- Sulfonylurea
Number analyzed (Participants) | 493 | 238
Percentage of HbA1c in the blood | -0.67 (0.044) | -0.79 (0.064)
Statistical Analysis 1: Comparison: Albiglutide 30 mg + Metformin +/- Sulfonylurea vs Insulin Glargine 10 Units + Metformin +/- Sulfonylurea; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.04 to 0.27]
Statistical Analysis 2: Comparison: Albiglutide 30 mg + Metformin +/- Sulfonylurea vs Insulin Glargine 10 Units + Metformin +/- Sulfonylurea; Test type: Non-Inferiority or Equivalence — To test whether the difference of least square means (albiglutide - insulin glargine) is equal to the pre-specified non-inferiority margin of 0.3%; p = 0.0086, t-test, 1 sided — p-value is for non-inferiority testing of albiglutide versus insulin glargine
Statistical Analysis 3: Comparison: Albiglutide 30 mg + Metformin +/- Sulfonylurea vs Insulin Glargine 10 Units + Metformin +/- Sulfonylurea; Test type: Superiority or Other; p = 0.1463, t-test, 2 sided — p-value is for superiority testing of albiglutide versus insulin glargine; The p-value is from a two-sided t-test to test whether the difference of least square means (albiglutide - insulin glargine) is equal to zero

2. Secondary Outcome: Change From Baseline in HbA1c at Week 156
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. Baseline HbA1c value is defined as the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. This analysis used observed HbA1c values, excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Time Frame: Baseline and Week 156
Population: ITT Population with observed values. Only those par. with a value at Baseline and at the specified visit were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c in the blood
Arm/Group | Albiglutide 30 mg + Metformin +/- Sulfonylurea | Insulin Glargine 10 Units + Metformin +/- Sulfonylurea
Number analyzed (Participants) | 123 | 88
Percentage of HbA1c in the blood | -0.83 (0.980) | -1.00 (0.922)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 52
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. The Baseline FPG value is the last non-missing value before the start of treatment. The LOCF method was used to impute missing post-Baseline FPG values. FPG values obtained after hyperglycemia rescue were treated as missing and replaced with pre-rescue values. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Based on ANCOVA: change = treatment + Baseline FPG + Baseline HbA1c category + prior myocardial infarction history + age category + region + current antidiabetic therapy.
Time Frame: Baseline and Week 52
Population: Intent-to-Treat (ITT) Population with LOCF. Only those participants with a value at Baseline and at the specified visit were analyzed. Values were carried forward for participants who were rescued or discontinued from active treatment before Week 52.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | Albiglutide 30 mg + Metformin +/- Sulfonylurea | Insulin Glargine 10 Units + Metformin +/- Sulfonylurea
Number analyzed (Participants) | 494 | 238
Millimoles per liter (mmol/L) | -0.87 (0.127) | -2.06 (0.184)

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 156
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. The Baseline FPG value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 156
Population: ITT Population with observed values. Only those par. with a value at Baseline and at the specified visit were analyzed. This analysis used observed FPG values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Albiglutide 30 mg + Metformin +/- Sulfonylurea | Insulin Glargine 10 Units + Metformin +/- Sulfonylurea
Number analyzed (Participants) | 119 | 86
Millimoles per liter (mmol/L) | -0.83 (2.803) | -2.19 (3.420)

5. Secondary Outcome: Number of Participants Who Achieved Clinically Meaningful HbA1c Response Levels of <6.5%, <7%, and <7.5% at Week 52
Description: The number of participants who achieved the HbA1c treatment goal (i.e., HbA1c response levels of <6.5%, <7%, and <7.5% at Week 52) were assessed.
Time Frame: Week 52
Population: ITT Population with LOCF. Only those participants with a value at Baseline and at the specified visit were analyzed. Values were carried forward for participants who were rescued or discontinued from active treatment before Week 52.
Measure: Number; unit: Participants
Arm/Group | Albiglutide 30 mg + Metformin +/- Sulfonylurea | Insulin Glargine 10 Units + Metformin +/- Sulfonylurea
Number analyzed (Participants) | 493 | 238
Participants
  HbA1c <6.5% | 54 | 25
  HbA1c <7% | 156 | 78
  HbA1c <7.5% | 268 | 135

6. Secondary Outcome: Number of Participants Who Achieved Clinically Meaningful HbA1c Response Levels of <6.5%, <7%, and <7.5% at Week 156
Description: The number of participants who achieved the HbA1c treatment goal (i.e., HbA1c response levels of <6.5%, <7%, and <7.5% at Week 156) were assessed.
Time Frame: Week 156
Population: ITT Population with observed values. Only those par. with a value at Baseline and at the specified visit were analyzed. This analysis used observed HbA1c values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide 30 mg + Metformin +/- Sulfonylurea | Insulin Glargine 10 Units + Metformin +/- Sulfonylurea
Number analyzed (Participants) | 123 | 88
Participants
  HbA1c <6.5% | 33 | 18
  HbA1c <7% | 59 | 46
  HbA1c <7.5% | 85 | 71

7. Secondary Outcome: Time to Hyperglycemia Rescue
Description: Participants who experienced persistent hyperglycemia (high blood glucose) could have qualified for hyperglycemia rescue. The conditions for hyperglycemia rescue were as follows: FPG >=280 milligrams/deciliter (mg/dL) between >=Week 2 and <Week 4; FPG >=250 mg/dL between >=Week 4 and <Week 12; HbA1c >=8.5% and a <=0.5% reduction from Baseline between >=Week 12 and <Week 24; HbA1c >=8.5% between >=Week 24 and <Week 48; HbA1c >=8.0% between >= Week 48 and <Week 156. Participants could have been rescued at any time on or after Week 2. Time to hyperglycemia rescue is defined as the time between the date of the first dose of study medication and the date of hyperglycemia rescue plus 1 day, or the time between the date of the first dose of study medication and the date of the last visit during the active treatment period plus 1 day for participants not requiring rescue. This time was divided by 7 to express the result in weeks.
Time Frame: From the start of study medication until the end of the treatment (up to Week 156)
Population: ITT Population. Only those participants with a value at Baseline and at the specified visit were analyzed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Albiglutide 30 mg + Metformin +/- Sulfonylurea | Insulin Glargine 10 Units + Metformin +/- Sulfonylurea
Number analyzed (Participants) | 496 | 239
Weeks | 107.57 [96.43 to 143.43] | NA [NA to NA] — There were too few events of hyperglycemia rescue (<50% of participants with events) to calculate the median and confidence interval.

8. Secondary Outcome: Change From Baseline in Body Weight at Week 52
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline weight minus the Baseline weight. The LOCF method was used to impute missing post-Baseline weight values. Weight values obtained after hyperglycemia rescue were treated as missing and replaced with prerescue values. Based on ANCOVA: change = treatment + Baseline weight + Baseline HbA1c category + prior myocardial infarction history + age category + region + current antidiabetic therapy.
Time Frame: Baseline and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Albiglutide 30 mg + Metformin +/- Sulfonylurea | Insulin Glargine 10 Units + Metformin +/- Sulfonylurea
Number analyzed (Participants) | 495 | 238
Kilograms | -1.05 (0.171) | 1.56 (0.247)

9. Secondary Outcome: Change From Baseline in Body Weight at Week 156
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline weight minus the Baseline weight.
Time Frame: Baseline and Week 156
Population: ITT Population with observed values. Only those participants who were available at the indicated time points were analyzed. This analysis used observed body weight values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Albiglutide 30 mg + Metformin +/- Sulfonylurea | Insulin Glargine 10 Units + Metformin +/- Sulfonylurea
Number analyzed (Participants) | 122 | 89
Kilograms | -3.47 (6.300) | 0.90 (4.890)

10. Secondary Outcome: Change From Baseline in Glucose Profile Measured by 24-hour Area Under Curve (AUC) at Week 52
Description: A 24-hour glucose profile was collected at Baseline and Week 52 at a subset of sites in a subset of participants per treatment group using the continuous glucose monitoring device. Glucose measurements were obtained at 5 minute increments in the 24-hour period. The area under the curve (AUC) was determined using the trapezoidal method on the measurements obtained during the first 24 hours of continuous monitoring. This analysis used observed values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed. The Baseline value is the last non-missing value before the start of treatment.
Time Frame: Baseline and Week 52
Population: Glucose Profile Substudy Population: all participants who participated in the 24-hour glucose profile substudy . Only those participants with a value at Baseline and Week 52 were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per hour per liter (mmol.h/L)
Arm/Group | Albiglutide 30 mg + Metformin +/- Sulfonylurea | Insulin Glargine 10 Units + Metformin +/- Sulfonylurea
Number analyzed (Participants) | 13 | 9
Millimoles per hour per liter (mmol.h/L) | 0.457 (2.9898) | -1.657 (1.9453)

11. Secondary Outcome: Albiglutide Plasma Concentrations at Week 8 and Week 24
Description: Albiglutide plasma concentration data was analyzed at Week 8 pre-dose, Week 8 post-dose, Week 24 pre-dose and Week 24 post-dose. All participants receiving albiglutide were initiated on a 30 mg weekly dosing regimen; however, beginning at Week 4, uptitration of albiglutide was allowed based on glycemic response. As such, albiglutide plasma concentrations achieved at each sampling time represent a mixed population of participants receiving either 30 mg or 50 mg weekly for various durations.
Time Frame: Weeks 8 and 24
Population: ITT population. Only those participants with a PK sample available for analysis at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Albiglutide 30 mg + Metformin +/- Sulfonylurea
Number analyzed (Participants) | 459
nanograms/milliliter (ng/mL)
  Week 8, Pre-dose, n=408 | 1642.83 (892.570)
  Week 8, Post-dose, n=398 | 1911.35 (966.180)
  Week 24, Pre-dose, n=416 | 2159.30 (1211.714)
  Week 24, Post-dose, n=401 | 2748.15 (1503.945)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs, defined as those events that had a start date on or after the first day of study medication and within 56 days after the end of study medication (up to Week 156), are reported.
Description: SAEs and non-serious AEs are reported for members of the Safety Population, comprised of all participants who received at least one dose of study treatment.
Arm/Group | Albiglutide 30 mg + Metformin +/- Sulfonylurea | Insulin Glargine 10 Units + Metformin +/- Sulfonylurea
Serious Adverse Events (participants affected / at risk) | 92/504 | 46/241
Other Adverse Events (participants affected / at risk) | 429/504 | 199/241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albiglutide 30 mg + Metformin +/- Sulfonylurea (N=504) | Insulin Glargine 10 Units + Metformin +/- Sulfonylurea (N=241)
Pneumonia (Infections and infestations) | 4 | 0
Bronchitis (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 1 | 2
Osteomyelitis (Infections and infestations) | 3 | 0
Diverticulitis (Infections and infestations) | 0 | 2
Lobar pneumonia (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Epiglottitis (Infections and infestations) | 1 | 0
Eye abscess (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Coronary artery disease (Cardiac disorders) | 5 | 2
Acute myocardial infarction (Cardiac disorders) | 3 | 2
Angina unstable (Cardiac disorders) | 2 | 3
Cardiac failure congestive (Cardiac disorders) | 2 | 2
Atrial fibrillation (Cardiac disorders) | 3 | 0
Myocardial infarction (Cardiac disorders) | 3 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Conduction disorder (Cardiac disorders) | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 5 | 4
Non-cardiac chest pain (General disorders) | 4 | 0
Death (General disorders) | 2 | 1
Device leakage (General disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Migraine (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Diabetic vascular disorder (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Cataract (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Albiglutide 30 mg + Metformin +/- Sulfonylurea (N=504) | Insulin Glargine 10 Units + Metformin +/- Sulfonylurea (N=241)
Upper respiratory tract infection (Infections and infestations) | 83 | 37
Nasopharyngitis (Infections and infestations) | 55 | 24
Sinusitis (Infections and infestations) | 50 | 23
Urinary tract infection (Infections and infestations) | 47 | 21
Bronchitis (Infections and infestations) | 44 | 27
Influenza (Infections and infestations) | 38 | 22
Gastroenteritis (Infections and infestations) | 19 | 6
Cellulitis (Infections and infestations) | 15 | 7
Pneumonia (Infections and infestations) | 12 | 5
Onychomycosis (Infections and infestations) | 12 | 2
Tooth abscess (Infections and infestations) | 11 | 4
Tinea pedis (Infections and infestations) | 11 | 1
Pharyngitis (Infections and infestations) | 10 | 6
Cystitis (Infections and infestations) | 5 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 187 | 117
Decreased appetite (Metabolism and nutrition disorders) | 14 | 4
Dyslipidaemia (Metabolism and nutrition disorders) | 12 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 50 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 37 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 | 17
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 21 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 17 | 19
Arthritis (Musculoskeletal and connective tissue disorders) | 11 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 6
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 4 | 6
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 67 | 18
Diarrhoea (Gastrointestinal disorders) | 55 | 19
Constipation (Gastrointestinal disorders) | 29 | 4
Vomiting (Gastrointestinal disorders) | 27 | 13
Dyspepsia (Gastrointestinal disorders) | 21 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 15 | 6
Abdominal pain (Gastrointestinal disorders) | 14 | 8
Toothache (Gastrointestinal disorders) | 5 | 5
Injection site reaction (General disorders) | 50 | 8
Oedema peripheral (General disorders) | 30 | 15
Injection site haematoma (General disorders) | 24 | 20
Fatigue (General disorders) | 21 | 3
Injection site erythema (General disorders) | 14 | 0
Chest pain (General disorders) | 5 | 8
Pyrexia (General disorders) | 5 | 7
Pain (General disorders) | 4 | 6
Headache (Nervous system disorders) | 46 | 20
Dizziness (Nervous system disorders) | 30 | 8
Diabetic neuropathy (Nervous system disorders) | 26 | 15
Carpal tunnel syndrome (Nervous system disorders) | 4 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 29
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 7
Asthma (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Hypertension (Vascular disorders) | 67 | 29
Anxiety (Psychiatric disorders) | 22 | 13
Depression (Psychiatric disorders) | 14 | 7
Insomnia (Psychiatric disorders) | 13 | 13
Cataract (Eye disorders) | 28 | 13
Diabetic retinopathy (Eye disorders) | 18 | 10
Rash (Skin and subcutaneous tissue disorders) | 15 | 10
Dermatitis contact (Skin and subcutaneous tissue disorders) | 9 | 5
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 5 | 5
Muscle strain (Injury, poisoning and procedural complications) | 10 | 8
Ligament sprain (Injury, poisoning and procedural complications) | 10 | 5
Contusion (Injury, poisoning and procedural complications) | 7 | 9
Anaemia (Blood and lymphatic system disorders) | 14 | 12
Vertigo (Ear and labyrinth disorders) | 11 | 6
Seasonal allergy (Immune system disorders) | 11 | 6
Weight increased (Investigations) | 6 | 5
Palpitations (Cardiac disorders) | 3 | 5
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.